CLINICAL TRIAL: NCT03406221
Title: Use of Mobile Technology to Improve the Performance of Community-Based Health Workers in Promoting Reproductive, Maternal, Newborn and Child Health and Nutrition Behaviors in Bihar, India: A Cluster Randomized Trial
Brief Title: Use of Mobile Technology by Community-Based Health Workers to Promote Maternal and Child Health in Bihar, India
Acronym: ICT-CCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Gary Darmstadt, Associate Dean for Maternal and Child Health, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-39719
Record Dates: First submitted 2017-10-23; First posted 2018-01-23 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Health; Pregnancy; Infant; Nutrition; Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental)
  Interventions: Behavioral: Information Communication Technology Continuum of Care Service
- Control Arm (Active Comparator)
  Interventions: Other: Control Condition

INTERVENTIONS:
Behavioral: Information Communication Technology Continuum of Care Service — Mobile phones were made available to community health workers in the intervention arms that integrated a comprehensive set of functions to assist them in their duties, including registration and tracking of beneficiaries, automated scheduling of home visits, provision of health information through videos, guided protocols for conducting home visits through checklists, a feature to track child immunizations, and supervisory tools.
  Arms: Intervention arm
Other: Control Condition — Standard of care
  Arms: Control Arm

SUMMARY:
This study is designed to evaluate the impact of use of mobile technology by community-based health workers on health-promoting behaviors among women related to reproductive, maternal, newborn and child health and nutrition in Bihar, India.

The intervention was funded by the Bill and Melinda Gates Foundation (BMGF) and in collaboration with CARE was implemented from 2012 to 2014. Health sub-centers in the catchment areas of four blocks (sub-districts) of the district of Saharsa were randomly assigned to treatment or control arms (35 sub-centers were assigned to each). Data were collected in the Intervention and Control areas from mothers of infants 0-12 months at baseline and at 2-year follow-up, to assess the intervention's effects on quality and quantity of FLW home visits, postnatal health behaviors, and among older infants/toddlers, complementary feeding and vaccination. Difference in difference analyses were used to assess outcome effects in this quasi experimental study.

The ICT-CCS intervention was implemented in areas where the BMGF-funded Ananya program (official title: Bihar Family Health Initiative) was also being implemented. Thus, the impact is of the [ICT-CCS intervention + Ananya] versus [Ananya alone]. The Ananya program was developed and implemented via a partnership of BMGF, CARE, and the Government of Bihar. The ultimate purpose of Ananya was to reduce maternal, newborn, and child mortality; fertility; and child undernutrition in Bihar, India. Ananya involved multi-level interventions designed to build front line health worker (FLW) capacities and reach to communities and households, as well as to strengthen public health facilities and quality of care to improve maternal and neonatal care and health behaviors, and thus survival. It was implemented from 2012 to 2014. Eight focal districts in western and central Bihar received Ananya, while 30 districts did not.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants 0-12 months residing in the catchment area of the subcenters

Exclusion Criteria:

-

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3112 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Receipt of two or more home visits from an FLW in the final trimester of pregnancy and delivery at a facility (versus home birth), using maternal survey response | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months; item created for Ananya Survey
Receipt of any postnatal home visits from an FLW (in the first 24 hours at home after delivery and in first month following delivery), using maternal survey response | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months; items created for Ananya Survey.
Any complementary feeding of solid or semisolid food for infants aged 6-11 months, using maternal survey response | 2 year follow-up
  A survey item was used to assess complementary feeding of infants as reported by mothers of infants aged 0-11 months; items created for Ananya Survey.
Immunizations | 2 year follow-up
  Receipt of DBT1 and DBT3 for infants 6-11 mo; receipt of DPT3 and measles vaccine for children 12-23 months; maternal receipt of at least 2 tetanus vaccines using immunization cards or maternal self-report if not card. Data from immunization cards or from self-reports when women did not have cards; approximately 50-60% of participants did not have immunization cards
Receipt of iron-folic acid tablets by month 4 and consumption of at least 90 tablets, using maternal survey response | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months; item created for Ananya Survey.
Clean Cord Care | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Kangaroo Mother Care (skin to skin care) | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Delayed Bath | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Initiation of Breastfeeding | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Nothing applied to cord or umbilicus | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Health worker placed child unclothed on mother's chest/abdomen in skin-to-skin contact | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
First bath delayed by two or more days | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months
Breastfed child within one hour of birth | 2 year follow-up
  Assessed via self-report from representative sample of mothers of children aged 0-11 months

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Carmichael SL, Mehta K, Raheel H, Srikantiah S, Chaudhuri I, Trehan S, Mohanty S, Borkum E, Mahapatra T, Weng Y, Kaimal R, Sivasankaran A, Sridharan S, Rotz D, Tarigopula UK, Bhattacharya D, Atmavilas Y, Munar W, Rangarajan A, Darmstadt GL; Ananya Study Group. Effects of team-based goals and non-monetary incentives on front-line health worker performance and maternal health behaviours: a cluster randomised controlled trial in Bihar, India. BMJ Glob Health. 2019 Aug 26;4(4):e001146. doi: 10.1136/bmjgh-2018-001146. eCollection 2019. PMID 31543982